CLINICAL TRIAL: NCT05236855
Title: Spectroscopy and Artificial Intelligence to Disrupt the Status Quo in Cervical Cancer
Brief Title: Spectroscopy and Artificial Intelligence to Disrupt the Status Quo in Cervical Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Cancer Society (CCS) (Other); Lancaster University (Other); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 1026741
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2021-08

CONDITIONS: Cervical Cancer; HPV
Keywords: Spectroscopy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine and cervical samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Women seen at the colposcopy clinic at Nova Scotia Health in Gynaecology-Oncology because of an abnormal cervical screen lab report
  Interventions: Diagnostic Test: Spectoscropy testing of urine specimen
- Control: Women seen at the General Gynaecology Clinic and the Izaak Walton Killam (IWK) Health Centre with a normal cervical screen lab report

INTERVENTIONS:
Diagnostic Test: Spectoscropy testing of urine specimen — Urine samples will be independently tested by I R Spectroscopy and those results are to be compared with standard testing procedures for HPV
  Groups: Intervention

SUMMARY:
Cervical cancer kills one woman every two minutes, 90% of these women are from low- and middle-income countries. Newly developed testing using biofluids has proven successful in identifying disease markers in, for example, brain cancers and endometrial cancers. Early studies have revealed that this technology is also showing potential for gynaecological cancers using validated human papillomavirus (HPV) test specimens. Urine samples, more easily collected, may make screening more accessible and acceptable to women. Spectroscopy is a portable and relatively simple technology; results are instant, reproducible and reliable. Once we confirm that spectroscopy has the ability to identify potential CIN 2+ by detecting HPV in urine, the test can be miniaturized and adapted to a point of care test. This will be more economical and logistically simpler than what is currently available; no consumables and pre-processing of samples are required. Women with abnormal cervical screening and women with normal screening as controls will be recruited, cervical and urine samples will be obtained. These will be tested for HPV DNA using standard methods and also by spectroscopy for HPV. These spectroscopy signals will be analyzed using artificial intelligence. The results will be compared to tissue samples obtained at colposcopy. This will allow evaluation of the new spectroscopy test. This preliminary study aims to prove the concept the spectroscopy as a simple, affordable screen can be used to radically change cervical cancer screening. Enabling a test that has point of care capabilities has huge implications for women in developed and more significantly in low-and middle-income countries, where cervical cytology and HPV testing have significant logistical problems. A non-invasive test will be preferred by many women. We believe spectroscopy will disrupt the status quo of 'no screening' in the low and middle income countries (LMICs), accelerate elimination of cervical cancer, and thus avert 15 million deaths in next 50 years.

DETAILED DESCRIPTION:
After obtaining informed consent, cervical and urine specimens will be obtained from all enrolled participants. Cervical biopsies in the disease group will be carried out at the providers' discretion per routine colposcopy protocols. Cervical specimens will be collected by the attending gynecologists and urine samples will be collected by the participants. Aliquots of urine and cervical samples will be tested for HPV DNA with cobas 4800 HPV test (Roche Diagnostics) serving as the gold standard at the Newfoundland Public Health Laboratory, St. John's, Newfoundland. The cobas test, however, identifies only two (types 16 and 18) of 14 high-risk HPV genotypes specifically. Therefore, a second set of aliquots will be tested at Seegene laboratory in Kitchener, Ontario to obtain complete genotype profile of all 14 high-risk genotypes as well as quantitative HPV results using Anyplex HPV DNA test (Seegene Inc), a next generation HPV test. Urine samples will also be independently tested by Infrared (IR) Spectroscopy and signals analyzed by Prof. Rehman's lab, Department of Engineering, Lancaster University, Lancaster United Kingdom (UK) to detect HPV. Spectroscopy results will be compared with HPV test results with genotypes to determine concordance between specimen types and between the testing technologies, with a special reference to urine testing. Biopsy confirmed CIN2+ will serve as the clinical endpoint to determine the sensitivity and specificity of urine spectroscopy testing in comparison with urine HPV testing; cervical HPV results will serve as the reference method. We are partnering with NSV-Tech a biotechnology company based in the US and India who have experience with artificial intelligence and cancer screening using tablet-based technology. Spectroscopy signals will be shared with NSV-Tech to develop artificial neural networks (ANN). The spectroscopy outputs linked to the ground-truth (biopsy confirmed abnormal cervical cells (CIN2)+ histology) will be used to develop ANN to improve diagnostic accuracy of this clinically relevant endpoint and remove subjectivity. The study relies on the ability for spectroscopy to detect HPV. The research team is confident this will be feasible. As noted, members of the research team are reviewing reference urine samples previously analyzed using standard HPV detection methods to confirm that spectroscopy is a viable option method. The control specimen collection and analysis uses standard methods. The data collection will take place in an academic colposcopy clinic with adequate patient volume and a proven track record in recruiting patients for such trials. The analysis of the spectroscopy in the UK of the spectroscopy, is in labs that have significant experience in assessing biological samples. The project's international collaboration is significant and brings together world class leaders in the prevention of cervical cancer who all have experience with novel technology and screening trials.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing standard HPV screening at the IWK Health Centre and Nova Scotia Health in Halifax, Nova Scotia, Canada

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women who undergo standard HPV screening
Study Population: Women undergoing standard HPV screening at the IWK Health Centre and Nova Scotia Health in Halifax, Nova Scotia, Canada
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Investigate the ability of spectroscopy to detect high risk HPV in urine | 18 months
  Confirm detection of HPV in urine using a new technique with I R Spectroscopy

SECONDARY OUTCOMES:
Measure the concordance between HPV detection by spectroscopy and by a validated HPV DNA test. | 18 months
  Comparison of standard HPV testing with a new method using I R Spectroscopy
Determine the sensitivity and specificity of urine spectroscopy for HPV | 18 months
  show that spectroscopy is non-inferior, clinically acceptable, to a validated HPV DNA test

REFERENCES:
- [Background] Paraskevaidi M, Morais CLM, Lima KMG, Snowden JS, Saxon JA, Richardson AMT, Jones M, Mann DMA, Allsop D, Martin-Hirsch PL, Martin FL. Differential diagnosis of Alzheimer's disease using spectrochemical analysis of blood. Proc Natl Acad Sci U S A. 2017 Sep 19;114(38):E7929-E7938. doi: 10.1073/pnas.1701517114. Epub 2017 Sep 5. PMID 28874525
- [Background] Sargent A, Fletcher S, Bray K, Kitchener HC, Crosbie EJ. Cross-sectional study of HPV testing in self-sampled urine and comparison with matched vaginal and cervical samples in women attending colposcopy for the management of abnormal cervical screening. BMJ Open. 2019 Apr 29;9(4):e025388. doi: 10.1136/bmjopen-2018-025388. PMID 31036707
- [Background] Pathak N, Dodds J, Zamora J, Khan K. Accuracy of urinary human papillomavirus testing for presence of cervical HPV: systematic review and meta-analysis. BMJ. 2014 Sep 16;349:g5264. doi: 10.1136/bmj.g5264. PMID 25232064
- [Background] Ogilvie GS, van Niekerk D, Krajden M, Smith LW, Cook D, Gondara L, Ceballos K, Quinlan D, Lee M, Martin RE, Gentile L, Peacock S, Stuart GCE, Franco EL, Coldman AJ. Effect of Screening With Primary Cervical HPV Testing vs Cytology Testing on High-grade Cervical Intraepithelial Neoplasia at 48 Months: The HPV FOCAL Randomized Clinical Trial. JAMA. 2018 Jul 3;320(1):43-52. doi: 10.1001/jama.2018.7464. PMID 29971397
- [Background] Mayrand MH, Duarte-Franco E, Rodrigues I, Walter SD, Hanley J, Ferenczy A, Ratnam S, Coutlee F, Franco EL; Canadian Cervical Cancer Screening Trial Study Group. Human papillomavirus DNA versus Papanicolaou screening tests for cervical cancer. N Engl J Med. 2007 Oct 18;357(16):1579-88. doi: 10.1056/NEJMoa071430. PMID 17942871
- [Background] Jackson R, Wang L, Jembere N, Murphy J, Kupets R. Why Do Women Get Cervical Cancer in an Organized Screening Program in Canada? J Low Genit Tract Dis. 2019 Jan;23(1):1-6. doi: 10.1097/LGT.0000000000000450. PMID 30489433
- [Background] Nishri ED, Sheppard AJ, Withrow DR, Marrett LD. Cancer survival among First Nations people of Ontario, Canada (1968-2007). Int J Cancer. 2015 Feb 1;136(3):639-45. doi: 10.1002/ijc.29024. Epub 2014 Jul 9. PMID 24923728
- [Background] McGahan CE, Linn K, Guno P, Johnson H, Coldman AJ, Spinelli JJ, Caron NR. Cancer in First Nations people living in British Columbia, Canada: an analysis of incidence and survival from 1993 to 2010. Cancer Causes Control. 2017 Oct;28(10):1105-1116. doi: 10.1007/s10552-017-0950-7. Epub 2017 Sep 8. PMID 28887646
- [Background] Brenner DR, Weir HK, Demers AA, Ellison LF, Louzado C, Shaw A, Turner D, Woods RR, Smith LM; Canadian Cancer Statistics Advisory Committee. Projected estimates of cancer in Canada in 2020. CMAJ. 2020 Mar 2;192(9):E199-E205. doi: 10.1503/cmaj.191292. Epub 2020 Mar 2. PMID 32122974
- [Background] Organization WH. Global strategy towards eliminating cervical cancer as a public health problem 2020. Available from: https://www.who.int/publications/m/item/draft-global-strategy-towards-eliminating-cervical-cancer-as-a-public-health-problem
- [Background] GLOBOCAN 2018: Estimated cancer incidence, mortality and prevalence worldwide in 2018: International Agency for Reserach on Cancer and World Health Organization. Available from: https://gco.iarc.fr/today/data/factsheets/cancers/23-Cervix-Uteri-fact-sheet.pdf.